## Informed Consent Form

Evaluation of Retinal Microvascular Change That May Develop in After Open Globe Injury

NCT05771467

November 27, 2023

Participant / Volunteer Protocol Number: 1. Information about the research:

a. Name of the Study Evaluation of Retinal Microvascular Change That May Develop in After Open Globe Injury

Purpose of the Research: As one of the most severe forms of ocular trauma, open-globe injury (OGI) causes significant vision loss. Timely and meticulous repair of these injuries can improve patient outcomes. After trauma, changes may occur in the non-trauma eye. Retinal and choroidal circulation may change as a result of adaptation mechanisms. In this study, we evaluated the vascular densities of the control group and post-traumatic non-trauma eye.

- b. Reason for the Research:
- (x) Scientific research () Thesis
- c. Estimated Duration of the Research: 6 months
- d. Number of Participants/Volunteers Expected to Participate in the Research: 50 patients / 50 controls
- e. Experimental Procedures to be Followed in the Research:

Participants' visual acuity, intraocular pressure, and anterior and posterior segment examinations will be performed. All examination procedures will be carried out in a non-contact and non-invasive manner.

2. Risks and Discomforts the Volunteer/Participant May Encounter During the Application:

I am aware that the procedures to be performed during the research described above may cause me the following risks and discomfort:

There is no risk

- 3. Expected Benefit of the Research for Volunteers/Participants: Detection of changes in posterior segment parameters of the healthy eye in traumatized patients.
- 4. Answering Questions on the Research Topic:

It will be sufficient to contact the person specified below to obtain information about possible side effects, risks and damages and my rights during the conduct of the research.

Name-Surname: ....... Phone: ...... 5. Compensation for Damages:

I was informed that if I were to be harmed because of my participation in this study, the necessary medical care would be provided by the responsible investigator, that I would be covered against any damage (including injury and death) that may occur due to the procedure performed, and that my expenses would be covered by ......

## 6. Research Expenses:

No fee will be charged from me or the social security institution to which I am affiliated for all transactions within the scope of the research.

- 7. Volunteering, Right to Refuse to Work and Withdrawal from Work, Dismissal from Work:
- a. I participate in the research voluntarily, without any pressure or coercion.
- b. I was informed that I had the right to refuse to participate in the study.
- c. I am aware that I can withdraw from this study at any time without giving any reason, provided that I notify the responsible researcher.
- 8. The researcher who is conducting the study or the supporting organization may exclude me from the scope of the study without my consent due to my negligence in fulfilling the requirements of the study program or depending on the research procedure.

## 9. Privacy:

The results of the study can be presented in scientific meetings or publications. However, in such cases my identity will be kept strictly confidential.

10. Consent to Participate in the Study:

I have read the text above, called Informed Consent Form, which shows the information that must be given to the volunteer / participant before the research, in my native language, or I have had it read to me. The content and meaning of this information was explained in written and verbal form. I was given the opportunity to ask all the questions that came to my mind and I received satisfactory answers to my questions. If I do not participate in the study or withdraw after participating, I will not waive any of my legal rights. Under these conditions, I agree to participate in this research voluntarily, without any pressure or coercion.

I received a signed copy of this text.

Name-Surname of the volunteer/participant: